CLINICAL TRIAL: NCT05146960
Title: The Effect of Evoked Temporal Summation in the Lateral Elbow Region on Cervical Muscle Endurance and Fatigue Characteristics
Brief Title: Relation Between Temporal Summation and Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BC-10785
Record Dates: First submitted 2021-10-29; First posted 2021-12-07 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Central Sensitisation; Elbow Pain; Fatigue
Keywords: motor performance; pain; temporal summation
MeSH Terms: conditions — Fatigue; Pain | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporal summation (Experimental): Temporal summation will be evoked in ECRL muscle origin, ECRB muscle belly, Brachioradialis. Pressure pain thresholds (PPTs) will be identified two times with a 30 s interval for each predetermined area. The average of two measurements will be used as a PPTs value. Temporal summation was induced two minutes after last PPTs was recorded. To evoke temporal summation at the lateral elbow, the probe will be applied with the pressure of the predefined PPT threshold at the rate of approximately 2 kg/s where it will be maintained for 1 s before being released with a 1 s interstimulus interval (ISI). This procedure will be repeated 10 times in each predetermined area. Pain intensity will be asked to participants at first, fifth and tenth pulse using a Visual Analog Scale range from "0 indicate no pain" to "10 most painful
  Interventions: Other: Temporal summation
- Placebo (Placebo Comparator): pressure pain threshold will be evaluated once in each predetermined region with a 30 second interval.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Temporal summation — Temporal summation will be evoked in each predetermined area
  Arms: Temporal summation
Other: Placebo — PPTs will be assessed once in each predetermined area
  Arms: Placebo

SUMMARY:
Central sensitization (CS) is a common feature in chronic musculoskeletal pain conditions including rheumatoid arthritis, chronic whiplash syndrome, fibromyalgia, temporomandibular joint disorders, low back pain and lateral elbow pain. CS is defined as "an amplification of neural signaling within the central nervous system that elicits pain hypersensitivity". Clinical signs are allodynia, hyperalgesia and widespread pain, originating from the enhanced activity of central nervous system to peripheral afferent input from unimodal and polymodal receptors.

CS not only induces abnormal pain processing, it may also lead to motor performance dysfunction in chronic pain population. CS induce cortical reorganization including changes in gray matter, cortical representation and cortical excitability both in motor and somatosensory cortex. This process ultimately generates sensorimotor conflict that described as a mismatch between motor intention and sensory feedback, and may directly effect on motor performance. The structural changes in basal ganglia and reduced GABAergic activity in the motor cortex contribute to the alteration of the motor performance. It has been known that CS and fatigue, another indicator of the motor performance, has a bidirectional effect and fatigue is predicted by CS, independently of the presence of pain. CS affect fatigue via causing disrupted reward process, increased effort and pain expactation.

The increased cervical spine hypersensitivity in patients with LEP even if there is no accompanied neck or upper limb pain may also indicate of the fatigue as pain does not always suggest an injury and biomechanical damage to a tissue does not always suggest that an individual will experience pain. If neck muscle fatigue is effected by central sensitization in patients with LEP, it can be important to develop therapeutic strategies to prevent neck muscle fatigue as there is a relationship between fatigue and increased risk of injury. Despite the fact that central sensitization effect on neck pain has been well documented in patients with LEP, its role on fatigue had not gain enough clinical and research attention. To know about central sensitization effect on motor performance can also be useful for determine subgroup of population who have central sensitization. However, it is unknown whether remote body endurance alteration occur in lateral elbow pain or not.

DETAILED DESCRIPTION:
EMG assessment Electrode Placement Before electrode placement, the skin will be cleaned with alcohol to reduce skin impedance.

Sternocleidomastoid Muscle (SCM) Electrode Placement Electrodes will be placed to the the sternal head of the SCM while participants were sitting in a erect position. A line will be drawn from the sternal notch to the mastoid process and marked at 1/3 of the distance from the sternal notch. Electrodes initially will placed adjacent to the this point with 20 mm apart and over the muscle belly based on the muscle palpation during manually resisted neck flexion contractions. This location is anticipated to place between the innervation zone and the tendon. In supine, the head will be placed in a neutral anatomic position that craniocervical and cervical spine is in a mid position. It will be ensured visually by examiner that cervical spine is in the neutral position which means from the middle of the subject's forehead to the middle of the chin is horizontal and a line bisecting the neck longitudinally is parallel to the treatment plinth. Participants will asked to completely relax in this position. For normalization, isometric neck flexor contraction will be carried out in supine position via applying manual resistance on frontal region by gradually increasing force that reached maximum force level in 2 second and then contracted maximally for 5 second. This procedure will be repeated 3 times with a 30 second time interval.

Upper Trapezius (UT) Muscle Electrode Placement Electrodes will be attached 20% laterally to the midpoint between the dorsal processes of C4 and the posterior lateral third of the clavicle. For normalization, manual resistance will be given neck extensor while participant lying in prone position. Contraction will be lasted 5 second for 3 times with 30 interval.

After electrode placement, a 5 seconds rest recording will be performed for eliminating basal noise from recording. During the endurance test, participants will asked not to cough, laugh or talk and head position will be controlled by inclinometer adapted to EMG system. Participants will be given 3 minutes resting time between neck flexor/extensor endurance tests for the experimental group.

Neck Flexor Endurance Test An examiner will place her hand under the occiput of the participant, while the participant is lying in supine position with the knees bend and the arms resting on the abdomen. Cranicervical flexion will be taught to the participants. For this, participants will asked to place tongue on roof of the mouth, with lips together and teeth slightly apart while cervical spine is in neutral position. Participants will not be allowed to open mouth during the test. Participants will be requested to perform gentle head nodding as if saying "yes" via sliding head in caudal and cephalic directions on the bed and concentrate feeling of back of the head. After learning of the craniocervical flexion, the participant will be requested to head off from the examiners hand (approximately 2.5 cm from the plint) vhile maintaining the craniocervical flexion and then sustain this position as long as possible. The holding time will be recorded with a stopwatch. The test will be ended once the participant is unable to hold their head in a correct position that chances occur more than 5 degree for more than one second, can no longer maintain craniocervical flexion or head position due to fatigue.

Neck Extensor Endurance Test Participants will be asked to lie in a prone position maintaining thoracal extension with a strap at the level of T6, arms in their side and head is end of the plinth. The subject's head and neck will be positioned in a comfortable neutral position with the chin retracted. 2 kg weight will be placed around the participants head. Participants will be asked to sustain this position as long as possible after removing support from the head. The test will be ended when the participant can no longer sustain a correct position or when the head position changes more than 5 degrees. The holding time will be recorded with a stopwatch.

Experimental group:

Experimental pain induction: Temporal Summation Then participants will be asked to seat in a comfortable position placing their volar faces of the tested dominant arm in elbow flexion on a table during the experiment. The tested area will be marked with a pen to apply every stimulus in the same place.

Temporal summation will be evoked in a predetermined area:

1. ECRL muscle origin: Distal humerus supracondylar ridge;
2. ECRB muscle belly: identified with resisted radial wrist flexion
3. Brachioradialis: 2 cm distal from in the middle of the line extend from lateral epicondyle to middle of the fossa cubiti via identifying resisted elbow flexion in 90° elbow flexion and wrist in neutral position Pressure pain thresholds (PPTs) will be identified two times with a 30 s interval for each predetermined area via applying circular probe in a perpendicular direction with an increasing pressure at a rate of approximately 1 kg/s. PPTs will be recorded when the sensation of the mechanical pressure stimulus changes into the first painful sensation. The average of two measurements will be used as a PPTs value. Temporal summation was induced two minutes after last PPTs was recorded. To evoke temporal summation at the lateral elbow, the probe will be applied with the pressure of the predefined PPT threshold at the rate of approximately 2 kg/s where it will be maintained for 1 s before being released with a 1 s interstimulus interval (ISI). This procedure will be repeated 10 times in each predetermined area. Pain intensity will be asked to participants at first, fifth and tenth pulse using a Visual Analog Scale range from "0 indicate no pain" to "10 most painful".

Placebo Group: After flexor and extensor endurance test, participants will be provided 20 minutes resting time. PPTs value will be evaluted once in each predetermined region with a 30 s interval.

Before PPTs assessment in predetermined area on lateral elbow, a familirisation session for the perceived PTTs by participants will be performed on palm of the non dominant arm for each group.

ELIGIBILITY:
Inclusion Criteria:

* To be healthy

Exclusion Criteria:

* have suffered pain at an intensity of more than 2/10 for more than 8 days in the preceding year;
* having had a pain condition in the last 6 months for which treatment was sought;
* have undergone surgery in the neck or elbow region in the preceding year;
* suffer major depression or psychiatric illness (diagnosed by a psychiatrist and being in medical or psychiatric treatment);
* be diagnosed with life threatening, metabolic, cardiovascular, neurologic, systemic diseases;
* be pregnant or have given birth in the preceding year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Sternocleidomastoid muscle normalized median frequency of the slope at 20 minutes | Baseline and minutes 20
  It shows fatigue characteristic of the muscle

SECONDARY OUTCOMES:
Change from baseline upper trapezius muscle normalized median frequency of the slope at 20 minutes | Baseline and minutes 20
  It shows fatigue characteristic of the muscle
Changes from baseline mean amplitude of the sternocleidomastoid muscle at 20 minutes | Baseline and minutes 20
  It shows fatigue characteristic of the muscle
Changes from baseline mean amplitude of the upper trapezius muscle at 20 minutes | Baseline and minutes 20
  It shows fatigue characteristic of the muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canli K, Palmans T, Meeus M, De Meulemeester K. Excitation of the bottom-up pathways has no effect on remote muscle fatigue in healthy participants. Exp Brain Res. 2024 Nov 27;243(1):2. doi: 10.1007/s00221-024-06958-w. PMID 39601827